CLINICAL TRIAL: NCT02584764
Title: Internet Supported Group Cognitive Behavior Therapy for Hoarding Disorder - A Pilot Study
Brief Title: Internet Supported Group Cognitive Behavior Therapy (CBT) for Hoarding Disorder (HD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Christian Rück, Associate Professor, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Hoarding Pilot
Record Dates: First submitted 2015-10-13; First posted 2015-10-23 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Hoarding Disorder
MeSH Terms: conditions — Hoarding Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CBT with Internet support (Experimental): 16 sessions of Cognitive behavior therapy in group with Internet support between group sessions
  Interventions: Behavioral: Cognitive behavior therapy; Behavioral: Internet support

INTERVENTIONS:
Behavioral: Cognitive behavior therapy
  Other Names: CBT
Behavioral: Internet support

SUMMARY:
The primary aim is to develop, and test the feasibility and efficacy of, a manual based, cognitive behaviour therapy (CBT) treatment for Hoarding Disorder (HD) delivered in a group format combined with an Internet support system. The investigators' secondary aim is to investigate the neurocognitive profile of the participants before and after treatment in order to explore if the treatment might have an impact on neurocognitive functioning and if certain neurocognitive profiles predict outcome.

For the primary aim, the investigators hypothesize that the treatment will be acceptable to participants and decrease symptoms of hoarding. Regarding the secondary aim, the investigators hypothesize that deficiencies in executive functioning, as measured with a neurocognitive battery, will reduce upon completion of treatment and that baseline executive function will be associated with treatment outcome.

ELIGIBILITY:
* Inclusion criteria:

  * Outpatients
  * Male or female
  * ≥ 18 years of age
  * Currently living in Stockholm county
  * Primary diagnosis of Hoarding Disorder according to DSM-5
  * Signed informed consent
  * Regular access to a computer with Internet and ability to use Internet
  * Access to a mobile phone
  * Able to participate in group sessions
* Exclusion criteria:

  * Current substance dependence or misuse
  * Life time bipolar disorder or psychosis
  * Severe self-rated depressive symptoms (score ≥ 35 on MADRS-S)
  * Suicidal ideation (score > 4 on item 9 in MADRS-S)
  * Psychotropic medication changes within two months prior to the treatment
  * Other current psychological treatment that could affect hoarding symptoms
  * Has received more than 10 CBT sessions for Hoarding Disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Saving Inventory - Revised (SI-R) | Change from baseline to treatment week 8,16, 3- and 12-month follow-up
  The SI-R is a 23-item self-report questionnaire. It assesses hoarding symptoms in 3 sub-scales: difficulty discarding, clutter and excessive acquisition.

SECONDARY OUTCOMES:
Hoarding Rating Scale - Self Report (HRS-SR) | Weekly change during treatment, weeks 1-15
  A 5-item self-report questionnaire assessing hoarding symptoms.
Saving Cognitions Inventory (SCI) | Change from baseline to treatment week 8,16, 3- and 12-month follow-up
  The questionnaire is a 24-item self-report questionnaire assessing beliefs and attitudes participants experience when trying to discard items. It is divided in 4 subscales:emotional attachment to objects, beliefs about objects as memory aids, responsibility for not wasting possessions, and the need for control over possessions.
Clutter Image Rating (CIR) | Change from baseline to treatment week 8,16, 3- and 12-month follow-up
  This scale consists of three sets of photographs each containing nine photos of a single room with varying levels of clutter. Study participants will select the photograph that best resembles his or her own home. The study investigators will also conduct blinded ratings of the same photos.
Global Assessment of Functioning (GAF) | Change from baseline to treatment week 8,16, 3- and 12-month follow-up
  A scale used to rate the social, occupational, and psychological functioning of the study participants.
Clinical global impression (CGI) | Change from baseline to treatment week 8,16, 3- and 12-month follow-up
  A 7 point scale to rate how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention.
EuroQol- 5 Dimension (EQ-5D) | Change from baseline to treatment week 8,16, 3- and 12-month follow-up
  A self-rating scale assessing quality of life i 5 dimensions.
Trimbos and Institute of Medical Technology Assessment Cost Questionnaire for Psychiatry (TIC-P) | Change from baseline to treatment week 8,16, 3- and 12-month follow-up
  In this questionnaire, study participants register their monthly health care consumption (e.g. GP visits) as well as time spent in informal health enhancing activities (e.g. self-help groups and informal care from friends). Additionally, work loss and work cutback both at work and in the domestic realm is measured.

OTHER OUTCOMES:
Hoarding disorder diagnosis | Change from baseline to treatment week 8,16, 3- and 12-month follow-up
  Presence of Hoarding Disorder according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5). Assessed by the investigators using the Structured Interview for Hoarding Disorder.
Comorbid psychiatric diagnoses | Change from baseline to treatment week 8,16, 3- and 12-month follow-up
  Presence of psychiatric diagnoses other than Hoarding Disorder. Assessed by the investigators using the M.I.N.I. International Neuropsychiatric Interview (M.I.N.I. 6.0).
Neuropsychological Test Battery (CANTAB) | Change from baseline to treatment week 16
  Cambridge Automated Neuropsychological Test Battery (CANTAB) will be used to test the study participants in 3 aspects of executive function: shifting and flexibility of attention, visuospatial working memory and response inhibition
Client Satisfaction Questionnaire - 8 (CSQ-8) | At treatment week 16
  An 8-item questionnaire measuring treatment satisfaction and acceptability.
Homework adherence | Weekly change during treatment, weeks 1-15
  Self-reported time spent on homework each week.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Rück, Assoc Prof, Principal Investigator — Karolinska Institutet
Locations (1):
- Psykiatri Nordväst, Stockholms Läns Sjukvårdsområde (SLSO), Stockholms Läns Landsting, Stockholm, Sweden